CLINICAL TRIAL: NCT00223054
Title: Polymorphism of the Cytochrome P450-system and the MDR-system in Renal Transplants Receiving the Immunosuppressive Drugs Tacrolimus, Sirolimus, Everolimus or Cyclosporine A
Brief Title: Polymorphism of the Cytochrome P450-system in Renal Transplants
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University of Kiel (Other)
Responsible Party: Lutz Renders, University of Kiel
Other Study IDs: 004
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2008-06

CONDITIONS: Function of Renal Transplant
Keywords: cyclosporin A; Tacrolimus; Everolimus; Sirolimus; Fluvastatin
MeSH Terms: interventions — Tacrolimus; Sirolimus; Everolimus; Cyclosporine

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA samples to analyze polymorphisms
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: tacrolimus — retrospective analyze of drug levels in comparison to polymorphism
Drug: sirolimus — retrospective of drug blood trough levels in comparison to polymorphism of enzymes of drug metabolism
Drug: everolimus — retrospective of drug blood trough levels in comparison to polymorphism of enzymes of drug metabolism
Drug: cyclosporin A — retrospective of drug blood trough levels in comparison to polymorphism of enzymes of drug metabolism

SUMMARY:
In this study the researchers want to investigate genetic polymorphisms of cytochrome 450 enzymes and the multiple drug resistance (MDR) gene in renal transplant patients to look for differences in dosing of immunosuppressive drugs (tacrolimus, sirolimus, everolimus, cyclosporine A).

All patients who receive one of these drugs can be included and drug blood trough levels, dosing and genetics are compared.

DETAILED DESCRIPTION:
Primary endpoint is the

1. serum creatinine in patients with and without polymorphysms
2. rate of rejections in patients with and without polymorphysms

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant patients receiving one or more of the following drugs:

  * tacrolimus
  * sirolimus
  * everolimus
  * cyclosporin A
  * fluvastatin
* Informed consent given by the patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patinets after kidney transplantation
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2005-03; Primary Completion 2006-06 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Renders, MD, Principal Investigator — University of Schleswig-Holstein, Campus Kiel, Department of Nephrology
Locations (1):
- University of Schleswig-Holstein, Campus Kiel, Department of Nephrology, Kiel, Germany

REFERENCES:
- [Result] Renders L, Frisman M, Ufer M, Mosyagin I, Haenisch S, Ott U, Caliebe A, Dechant M, Braun F, Kunzendorf U, Cascorbi I. CYP3A5 genotype markedly influences the pharmacokinetics of tacrolimus and sirolimus in kidney transplant recipients. Clin Pharmacol Ther. 2007 Feb;81(2):228-34. doi: 10.1038/sj.clpt.6100039. Epub 2006 Dec 27. PMID 17192769